CLINICAL TRIAL: NCT04852198
Title: A Study on Safety and Efficacy Comparing 150cm One Anastomosis Gastric Bypass With 150cm Biliopancreatic Limb Roux-en-Y Gastric Bypass (Roux-en-WHY?): An Open Label, Multicentre Non-inferiority Randomized Controlled Trial
Brief Title: Comparing 150cm OAGB With 150cm Biliopancreatic Limb RYGB. A Non-inferiority Trial
Acronym: Roux-en-WHY?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Flevoziekenhuis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FZ 20/22; NL74137.018.20 (Other: CCMO)
Record Dates: First submitted 2020-10-06; First posted 2021-04-21 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Bariatric Surgery Candidate; Obesity; Obesity, Morbid
MeSH Terms: conditions — Obesity; Obesity, Morbid

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with 2 groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OAGB (Active Comparator): 149 patients receiving one anastomosis gastric bypass (OAGB) with a Biliopancreatic-limb of 150cm
  Interventions: Procedure: OAGB
- RYGB (Active Comparator): 149 patients receiving Roux-en-Y gastric bypass (RYGB) with a Biliopancreatic-limb of 150cm
  Interventions: Procedure: RYGB

INTERVENTIONS:
Procedure: OAGB — Simplified gastric bypass procedure
  Other Names: Mini gastric bypass; Omega loop gastric bypass
  Arms: OAGB
Procedure: RYGB — Roux-en-Y gastric bypass. Standard procedure in the Netherlands
  Arms: RYGB

SUMMARY:
The purpose of this study is to assess the safety and efficiency of OAGB compared to RYGB

DETAILED DESCRIPTION:
Rationale: to compare two different types of gastric bypass operations on surgical outcome.

Objective: to compare two established procedures in order to find the optimal procedure in terms of weight loss and metabolic control that is associated with the fewest side-effects and complications, and decreased invasiveness.

Study design: A multicentre, open label, non-inferiority randomized controlled trial Study population: Patients are eligible for inclusion if their body-mass index (BMI) was 40 kg/m2 or higher, or 35 kg/m2 or higher with the presence of at least one comorbidity (type 2 diabetes, high blood pressure, obstructive sleep apnoea, dyslipidaemia, osteoarthritis of the hip or knee) and a positive evaluation by our bariatric multidisciplinary team (BMDT) and are aged 18-65.

Intervention: Group 1: One Anastomosis Gastric Bypass with 150cm biliopancreatic limb. Group 2: Roux-en-Y gastric bypass with biliopancreatic limb of 150cm and 75cm alimentary limb.

Main study parameters/endpoints:

Primary endpoint:

% Excess BMI loss at two years

Secondary endpoints:

Metabolic status Nutritional status Comorbidity remission QOL Complications or serious adverse events (SAE's)

ELIGIBILITY:
Inclusion Criteria:

* body-mass index (BMI) of 40 kg/m2 or higher, or 35 kg/m2 or higher with the presence of at least one comorbidity (type 2 diabetes, high blood pressure, obstructive sleep apnoea, dyslipidaemia, osteoarthritis of the hip or knee)
* a positive evaluation by our BMDT

Exclusion Criteria:

* Presence of H. Pylori, resistant to eradication therapy
* chronic diarrhoea
* history of previous bariatric or extensive abdominal surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Estimated)
Dates: Start 2021-12-13 (Actual); Primary Completion 2027-06-13 (Estimated); Study Completion 2029-11-01 (Estimated)

PRIMARY OUTCOMES:
Percentage excess BMI loss at 2 years (%EBMIL) | 2 years
  Percentage excess BMI loss after 2 years of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Stef JM Smeets, MD PhD, Principal Investigator — Flevoziekenhuis
Locations (2):
- Netherlands (2):
  - Flevoziekenhuis, Almere Stad
  - OLVG, Amsterdam

IPD SHARING:
Plan to Share IPD: No